# CONSENT TO TAKE PART IN A CLINICAL RESEARCH STUDY AND AUTHORIZATION TO DISCLOSE HEALTH INFORMATION

Study Title: "A Phase 1b Study of CG0070 Combined with Nivolumab in

Cisplatin Ineligible Patients with Muscle Invasive Bladder

Cancer (MIBC)"

Protocol Number: CORE-002

Sponsor: Moffitt Cancer Center

Principal Roger Li, MD Investigator:

(Study Doctor)

Telephone: 813-745-8343

(24 hour number) (800) 456-3434 (813) 745-8000

Address: Moffitt Cancer Center

12902 Magnolia Drive Tampa, FL 33612

**Moffitt Cancer Center – McKinley Campus** 

10920 N. McKinley Drive

Tampa, FL 33612

You are being asked to take part in a clinical trial. A clinical trial is a type of study that involves research. Clinical trials only include participants who choose to take part. This document, called an informed consent, provides information to help you make an informed decision as to whether or not you wish to take part in the study.

The goal of this clinical research study is to find out if CG0070 along with Nivolumab is effective in treating your cancer condition. We are asking you to take part in this research study because you have bladder cancer that has invaded the muscular wall and you are not able to take the standard treatment of cisplatin. You have already been diagnosed with bladder cancer and you will have surgery after the study treatment.

Before you can start the study, the study doctor or study staff will talk to you about the study. If you agree to participate, you have to sign and date this form before the study doctor or study staff can begin the first part of the study called a screening period (for a period of up to 14 days)



to see if you qualify to be in the study treatment phase of the study. Your study doctor will determine your eligibility to participate in the study. If you qualify to continue in the study you will undergo a study treatment visit. This will involve administration of the investigational drug along with other study procedures which are later described in detail in this document. After the study treatment visit, you will have an end of study treatment/follow-up visit which involves evaluating your health condition by routine clinic examination and procedures, later described in detail. Your regular medical care might include some of the study tests and procedures. The study doctor or a member of the study staff can answer any questions you may have about which tests and procedures are not part of your regular medical care.

About 18 local participants will be invited to take part in this research. The total number of participants across all sites will be around 30.

Your participation is voluntary, and you may stop your participation at any time. There will be no penalties, loss of benefits or opportunities if you do not participate or decide to stop once you start. Alternatives to participating in the study are later described in this document.

We do not know if you will receive any benefit from your participation. There is no cost to participate. You will not be compensated for your participation. The most common and most serious risks that may be related to taking part in this research are dysuria, diarrhea, fatigue, itching and rash. Additional risks are described later in this consent form.

Any new important information that is discovered during the study and which may influence your willingness to continue participation in the study will be provided to you.

Even if we publish the findings from this study, we will keep your study information private and confidential. Anyone with the authority to look at your records must keep them confidential.

If you are interested in learning more about this study, please continue reading the information below.

#### WHAT IS THIS STUDY ABOUT?

You are being asked to participate in this research study because you have been diagnosed with bladder cancer that has invaded the muscular wall. This is called muscle invasive bladder cancer (MIBC). You may have been treated with other intravesical agents for your cancer as well.

The main purpose of this study is to find out whether CG0070, DDM, and nivolumab are safe when given together, whether your tumor disappears after study treatment (called a complete response), and if you have a complete response, to monitor how long the response lasts.

The agents (study drugs) as used in the study are experimental. There is no guarantee that they will improve or stabilize your cancer. In fact, these agents may make you worse. The experimental agents (study drugs) being studied are called **CG0070**, **DDM**, **Nivolumab**.

MCC #:20575

**CG0070** is a virus (called Adenovirus, serotype 5) that has been altered in a laboratory (genetically modified) to infect and destroy cancer cells and release a protein called GM-CSF along with an E2F promoter that plays a role in the defense system fighting cancer. As of January 2022, over 162 participants have received CG0070 in over 500 total study treatments. CG0070 has not been approved by any regulatory agency, including the U.S. Food and Drug Administration (FDA), for sale anywhere in the world.

**DDM** (also known as n-dodecyl-B-D-maltoside) is a sugar based non-ionic mild detergent that acts like solubilizing agent to increase the passing of CG0070 through of mucous membrane of the bladder. It has been used as a food additive, as an intravenous (IV), and as an intranasal component in other drugs, some approved by the United States FDA.

**Nivolumab** is an anti-PD-1 (programmed cell death) antibody. It works by attaching to and blocking a molecule called PD-1. PD-1 is a protein that is present on different types of cells in your immune system and controls parts of your immune system by shutting it down. Antibodies that block PD-1 can potentially prevent PD-1 from shutting down the immune system, thus allowing it to recognize and help your body destroy the cancer cells.

Nivolumab has not been approved by the U.S Food and Drug Administration (FDA) to be used for muscle invasive bladder cancer prior to definitive surgical treatment (in the "neoadjuvant setting"), so it is being considered "investigational" for use in this study. An investigational drug is a drug that is being tested and is not approved for sale in the United States by the U.S. Food and Drug Administration (FDA).

OPDIVO® (nivolumab) is approved by the FDA for the treatment of multiple other tumor types and is available to be prescribed for patients with those diseases.

#### WHAT WILL HAPPEN DURING THIS STUDY?

This consent form will describe the 3 distinct phases of participation: Screening Phase, Study Treatment Phase, and Follow-Up Phase. The Screening Phase will last up to 28 days. The Study Treatment Phase can continue for up to 24 months from the start of study treatment unless your cancer gets worse or recurs. The Follow-Up Phase will last for up to 4 years from the start of study. You will not be scheduled to return to the clinic/hospital for the study during the Follow-Up Phase, but you will be contacted about every 12 weeks.

# Screening:

Your study doctor will complete the following procedures to determine if you are eligible to participate in the study. These tests or procedures include:

- 1. Signing and dating this informed consent document
- 2. Providing your medical and bladder cancer history, including any previous treatments vou received
- 3. Providing information on any medications you are currently taking or take occasionally
- 4. Physical examination including height, weight, and vital signs
- 5. Blood (approximately 1 tablespoon or 15 mL) and urine (approximately 1.5 tablespoon or 20 mL) tests to determine organ function

- 6. Urine Cytology (urine test) and Cystoscopy (bladder scope) to determine disease status
- 7. Pregnancy test (if you are a woman who is able to become pregnant)
- 8. Transurethral resection of bladder tumor (TURBT) to remove any residual tumor tissue using cytoscopy prior to beginning the trial (this will only be performed if you have not had one done within 12 weeks and if you have disease to remove)
- 9. Electrocardiogram (ECG) to look at the electrical activity of the heart.
- 10. Computerized tomography (CT) Urogram which is an imaging exam used to evaluate your urinary tract or magnetic resonance urography (MRU) to rule out any disease beyond the bladder

# **Study Treatment**:

Once your study doctor determines that you are eligible to participate in the study, you will be required to attend in-clinic study visits and have periodic evaluations to determine the safety and effectiveness of the combined CG0070, DDM, and nivolumab study treatment, as described in the Study Calendar at the end of this document. These tests or procedures include:

- 1. Collecting information on any medications you are currently taking or take occasionally
- 2. Physical examination including weight and vital signs
- 3. Blood (approximately 1 tablespoon or 15 mL) and urine (approximately less than 1.5 tablespoon or 20 mL) tests to determine organ function
- 4. Urine Cytology and CT scans to determine disease status
- 5. Biopsy, if applicable
- 6. Pregnancy test (if you are a woman who is able to become pregnant)
- 7. ECG

#### STUDY DRUG ADMINISTRATION

#### **Intravesical Procedure**

**CG0070** and **DDM** will be given by intravesical therapy, meaning that these agents will be put into your bladder using a catheter. At least 4 hours before study treatment you will need to avoid caffeinated beverages and minimize fluid intake. Your study doctor will explain what this means in more detail.

At the start of the intravesical procedure, you will be asked to empty your bladder completely, and then a urinary catheter will be installed in a procedure called a urinary catheterization. Your study doctor will then start the intravesical instillation procedure (administering study drug into the bladder). You will receive an initial bladder wash with 100 mL (about 6.5 tablespoons) of normal saline, followed by a second bladder wash of 75 mL (about 4.5 tablespoons) of DDM and your bladder will be emptied again. The study doctor will then infuse 100 mL of DDM into the bladder and it will stay in the bladder for 15 minutes. After 15 minutes, the fluid in the bladder will be removed and you will receive a third bladder wash with 100 mL of normal saline. The study doctor will then infuse the 100 mL of CG0070 mixed in normal saline into the bladder and it will stay in the bladder for 1 hour. The fluid in the bladder will be removed after 1 hour.

MCC #:20575

At the end of each intravesical study treatment, you will be asked to stay at the study center for at least 1 hour. Your study doctor may decide to observe you for longer depending on your signs and symptoms. This is mainly to monitor your conditions for any potential study treatment related adverse event. You may receive additional examination and tests for the safety assessment ordered by your study doctor.

Before being discharged after the study treatment, you will be educated by the study team on proper site care at home, hand hygiene and cough etiquette, and to avoid direct close contact with people who are potentially at higher risk from exposure.

#### **CG0070 and DDM Administration**

CG0070 and DDM will first be given as part of weekly study treatments for 6 weeks (Weeks 1, 2, 3, 4, 5, and 6).

#### **Nivolumab Administration**

Nivolumab will be administered by intravenous (IV) infusion, meaning the study drug is a solution given through a vein, on week 2 and week 6. A pump will be used to ensure the correct amount of study drug is given over the proper amount of time. The nivolumab infusions will take about 30 minutes. Nivolumab infusion will be followed by at least a 2 hour rest before CG0070 intravesical infusion is given.

The duration of your stay at the study site after the first infusion of nivolumab would be dependent on the hospital standards and the number of study procedures to be completed before, during and after infusion of study drug. The study doctor will inform you about the duration of your stay at the site in more details if needed.

# Follow-Up:

Once you finish study treatment and until you withdraw your consent, you will have routine follow up visits post-surgery at approximately every 3 months for up to two years in the absence of disease progression. At each visit, history, physical, laboratory workup, and imaging will be performed to evaluate for oncologic (tumor) and functional outcomes.

In addition, you will be contacted to collect information about any side effects you may have experienced after coming off study treatment with CG0070, DDM, and nivolumab for up to 100 days following your last study treatment.

# **Routine Procedures**

The following tests will be done as part of this study. Some of these tests may be done as part of your standard care and may not need to be repeated for the study, some of these tests may be done more frequently than if you were not taking part in this study, and some may be done solely for the study. If the results show that you are not able to continue participating, your study doctor will let you know.

 Physical examination, weight, height, and an assessment of your ability to care for yourself, called an ECOG performance status

- Vitals (blood pressure, heart rate and temperature)
- Routine blood tests to look at how well your bone marrow, liver, kidneys and thyroid
  gland are functioning and to look at the time it takes for your blood to clot. If you are a
  woman who can have a child, a pregnancy test will be performed periodically. These
  tests are performed at your study center and will be kept in your medical record.
- Electrocardiogram (ECG) electrical currents generated by the heart are recorded.
- Urine sample collection to look for abnormal cells in the urine
- Cystoscopy to examine the lining of your bladder and the tube (called urethra) that carries urine out of your body.
- Biopsy of pelvic lymph nodes to take samples of the tumor tissue from potentially affected lymph nodes
- Computerized Tomography (CT) Urogram or Magnetic Resonance Urography (MRU) to rule out any disease beyond the bladder,
- Transurethral Resection of Bladder Tumor (TURBT) to remove bladder tumor from the bladder wall.
- Radical Cystectomy to remove the bladder, the prostate, the seminal vesicles (sperm sacs), and, if necessary, the urethra.

#### Urinary Tract Evaluation

Before the study treatment, your study doctor will ask you to complete a series of examinations and scan tests to evaluate the urinary tract condition. Your study doctor will either perform a Computerized Tomography (CT) Urogram or Magnetic Resonance Urography (MRU) to rule out any disease beyond the bladder at the beginning of the study and every 3-months postoperatively on the study. However, if you have done the scan within 8 weeks of Day 1, you will not be asked to repeat the test.

# Urine Sample Collection

The researchers doing this study are interested in doing research on urine samples to better understand the nature of cancer in general and the study drugs passing that may be found in the urine particularly. The researcher will conduct a test, called Urine Cytology, looking for the abnormal cells in the urine during the study treatment period.

You will be asked to collect a sample of 2-4 tablespoons or 30–60 mL of urine "mid-stream" into a clean container, any excess urine should be voided into the toilet. The collection of urine samples is a necessary part of this study.

MCC #:20575

## Study-Specific (Non-Routine) Procedures

In addition to the tests that we will conduct to determine whether you are having side effects or if you are responding to the study therapy, we will also collect samples and perform tests for purposes of research only. Some of these tests may be optional and others may be required in order to participate in the study. These tests include:

- Blood, saliva, and urine tests to study how CG0070 and nivolumab act within the body and to study any changes to the immune system will be collected.
- Tumor biopsies: a procedure to remove pieces of tissue or a sample of cells from several areas within your bladder so that it can be analyzed in a laboratory and is used to diagnose or evaluate the cancer. You will be required to have a biopsy at least once: before you start study treatment, unless a biopsy was completed recently. If there is disease remaining at 9 weeks prior to cystectomy, an optional biopsy may be taken.
- Genetic testing Your tissue will help us study how genes might play a role in cancer and your response to CG0070 and nivolumab. The testing will be limited to genes that are not known to cause diseases; therefore, we will not share the results of these research tests with you.

#### **HOW WILL MY BLOOD/TISSUE SAMPLES BE USED?**

In addition to the procedures outlined above, we are asking you to allow us to obtain and store samples of your blood, tissue and urine collectively referred to as "tissue" for use in future research. These samples may be used for research on your disease or condition and others to assist in the development of new treatments.

If a biopsy was performed for entry into this clinical trial, your biopsy specimen will be retained in accordance with the current hospital or clinic policy, or local requirements. Future research on blood, urine and biopsy samples may be conducted by Moffitt, CG Oncology or 3<sup>rd</sup> parties. Any samples stored for future research will be de-identified, meaning personal information which could be used to identify you will be removed. Instead all samples will be given a unique code number assigned to you. We will not release the code that links your sample to your personal identifying information for any reason.

These research samples (blood, urine and biopsy) will be collected and analyzed in order to better understand the cancer and study treatment, including:

- How much CG0070 is present in your blood and urine and how long it remains in your blood and urine.
- How the drugs CG0070 and nivolumab work in the body.
- How your body reacts to CG0070 and nivolumab
- What makes some people respond better to the drug or drugs.

Research samples will be stored for 10 years and will be destroyed at the end of the storage period. The information gathered on this trial will be used by researchers from Moffitt Cancer

Center, CG Oncology, and 3<sup>rd</sup> parties that, after a thorough review and approval process, will be allowed to use these samples for the research purposes described in this consent form.

Reports about any research done with your samples will not be given to you or your study doctor. These reports will not be put in your medical records. The research using your samples will not affect your care.

You have the right to withdraw your consent to use/store your blood, urine and biopsy samples (including requesting destruction of the sample) as long as the link to your identity is unbroken, and without explaining the reasons for your decision. If you no longer want your blood, urine and biopsy samples to be used in this research, you should tell your study doctor. Your study doctor will notify the Sponsor, who will ensure that the samples are destroyed. If tests have already been done on your samples it will not be possible to withdraw your permission for those tests; however, no further testing will be done. However, if you withdraw your consent for future testing on these samples, you may be excluded from all future study visits sponsored by CG Oncology.

#### WHO IS PAYING FOR THIS STUDY?

A company called Cold Genesys Inc., the sponsor of the study, is paying for this study.

# WILL IT COST ANYTHING TO BE IN THIS STUDY?

You and/or your insurance company will be financially responsible for hospital inpatient, outpatient and follow-up visits that would normally or routinely occur in the management of your disease. Inpatient and outpatient visits could include charges for treatments, medications, physician visits, laboratory tests and procedures. You and /or your insurance company will be responsible for paying for the charges which are considered routine, since you would have received these services even if you were not participating in this study. You will be responsible for any costs not covered by your insurance company, including deductibles, co-payments and all out-of-pocket expenses. Before you agree to be in this study, you should contact your health insurer to see if your plan will cover the costs required as part of your participation.

You and/or your insurance company will not be responsible for paying for study related items and services that are specifically required for this research study and are not considered part of the routine management of your disease, if these procedures are performed at Moffitt Cancer Center.

During your participation in this study, CG Oncology, Inc. will be responsible for providing the study drugs, Nivolumab, CG0070 and DDM at no additional charge to you. You and/or your insurance company will be responsible for the charges related to the administration of the study drugs.

If you would like more information on the costs of being on this study or have other insurance related questions then please let your clinical trial coordinator know or contact our Business Office at 813-745-8422.

MCC #:20575

**Medicare Advantage:** If you are in Medicare Advantage (Medicare managed care plan), you should contact someone at your plan before you start a clinical trial. They can provide more information about additional costs you could incur from participating in clinical trials.

#### WILL BEING IN THIS STUDY HELP ME?

You may benefit as a result of your participation in this study. There is, however, no guarantee that you will benefit from your participation in this study. Information learned from the study may help other people in the future.

#### ARE THERE RISKS TO ME IF I AM IN THIS STUDY?

If you take part in this study, you are at risk for the side effects outlined below. You should talk to your study doctor about these side effects in case they happen. There also may be other side effects and sometimes serious side effects that are not yet known. Many side effects go away shortly after study treatments are stopped, but side effects could last a long time or could last forever. The side effects may range from mild to life-threatening. Your study doctor may give you other drugs to make side effects less serious and less uncomfortable.

Unknown and potentially life-threatening side effects could occur, or your condition could worsen. The study treatment may not be better than radical cystectomy alone; and the combination of the 3 study agents may result in worse or unknown side effects. Should any side effects or other reactions occur while in this study, notify your study doctor immediately.

If you experience side effects that require treatment between regular clinic/hospital visits, it is important that you make every effort to return to the clinic/hospital where CG0070 and nivolumab was given. Because CG0070 and nivolumab are experimental drugs and are only used in clinics/hospitals involved in research studies, any serious side effects of the drug may be best treated by these clinics/hospitals. If you need immediate treatment and are unable to return to the treatment clinic/hospital, you should go to the nearest emergency department and your study doctor should be contacted as soon as possible.

# **Accidental Transmission**

CG0070 is made from adenovirus. In nature, adenoviruses can cause flu-like, respiratory, and gastrointestinal symptoms. CG0070 has been weakened in a laboratory, but it still may be possible that the virus could be transmitted accidentally. You will be given a Patient Instruction Form with information on precautions to be followed while you are receiving the study treatment. These precautions are for the safety of other people around you that you may have close physical or direct contact with and are necessary so that you do not accidentally give them the virus. Please refer to this information sheet to minimize the risk of exposure to virus for any high-risk individuals that you might come in contact with should these symptoms occur.

MCC #:20575

#### HERE ARE THE KNOWN SIDE EFFECTS THAT COULD HAPPEN WITH CG0070

As of January 2022, approximately 162 participants with bladder cancer received CG0070. The majority of the side effects occurred to date were mild-to-moderate local genitourinary symptoms. After receiving CG0070 study treatment, side effects might occur relatively acutely, starting and resolving within a few days after the initial study treatment. Your study doctor will evaluate and decide on the treatment that includes supportive care measures.

If receiving CG0070, it is expected that your immune system will remove CG0070 from your body within approximately 30 days. However, because CG0070 is a living virus, it is possible that the virus may stay in your body for a longer period of time and cause other complications that are unknown.

In the extremely unlikely case that you develop a serious reaction and your study doctor thinks it is related to receiving CG0070, there are medications you may be offered that could help. Your study doctor will be responsible for treating you with one or more of these medications, if needed.

CG0070 and nivolumab have not been administered together before and while both drugs have shown to have similar side effects, it is not known if the combination of both drugs may lead to an increased severity of known side effects or may lead to additional side effects related to immune system activation.

The most common side effects related to CG0070 study treatment observed are described below.

**VERY COMMON:** In 100 people, may occur in 20 people or more:

Dysuria - painful urination

**COMMON:** In 100 people, 5 to 20 may have the following

•

- Sudden urgency to urinate that may be uncomfortable or embarrassing
- Hematuria blood in your urine
- Fatigue tiredness
- Bladder spasm (painful bladder camps)
- Urine abnormality
- Nocturia- waking up more than one time during the night to pass urine

**UNCOMMON:** In 100 people, 1 to 5 may have the following:

- Influenza like illness (flu like symptoms)
- Bladder discomfort
- Myalgia muscle pain
- Urinary Tract Infection
- Abdominal pain
- Arthralgia pain in the joint
- Influenza
- Headache
- Incontinence- lack of voluntary control over urination

MCC #:20575

- Nausea
- Bleeding from urinary system
- Hot Flush feeling of intense warmth
- Hypertension high blood pressure
- Urinary Tract and Urethral Pain pain in the urethra (the tube that passes from the bladder to the outside of the body
- Polyuria increase urination during the day
- Chills
- Malaise general feeling of discomfort, illness, or uneasiness
- Fever

#### **Possible Side Effects of Nivolumab**

Nivolumab may cause one or more of the side effects listed below. This information is based on data from cancer participants in other clinical trials with nivolumab. In addition, there may be side effects that are not yet known that may occur. You should tell your study doctor or study nurse right away about any possible side effects you experience.

Nivolumab may worsen any side effects that you may experience from your radiation therapy as well as any side effects that you may have experienced from your previous chemotherapy.

# **VERY COMMON**: may affect more than 1 in 10 people

- Diarrhea
- Fatigue tiredness
- Itchina
- Rash

# **COMMON**: greater than or equal to 1 in 100 to less than 1 in 10

- Abdominal (stomach) pain
- Alkaline phosphatase increased- lab test result associated with liver or bone abnormalities
- Allergic reaction/hypersensitivity
- ALT increased- lab test result associated with abnormal liver function
- Amylase increased- lab test result associated with pancreas inflammation
- AST increased- lab test result associated with abnormal liver function
- Bilirubin (liver function blood test) increased
- Chills
- Constipation
- Cough
- Creatinine increased- lab test result associated with decreased kidney function
- Decreased appetite
- Dizziness or vertigo -feeling off balance which can lead to dizziness
- Dry mouth
- Dry skin

- Fever
- Headache
- Increased blood sugar
- Inflammation of the colon
- Inflammation of the mouth
- Joint pain or stiffness
- Lipase increased- lab test result associated with pancreas inflammation
- Loss of color (pigment) from areas of skin
- Low levels of sodium in the blood
- Low platelet counts (thrombocytopenia): this may increase your risk for skin bruising, nose bleeds, and bleeding from the gums
- Low red blood cell counts (anemia): this may make you feel weak and tired
- Lung inflammation -pneumonitis see details below
- Nausea (upset stomach)
- Pain in the muscles, bones, ligaments, tendons, and nerves
- Reaction related to infusion of the medicine. The symptoms may include but not limited to fever, rash, pain, swelling
- Shortness of breath
- Swelling, including face, arms, and legs (edema)
- Thyroid gland function decreased or may be increased; increased thyroid stimulating hormone a lab test result associated with abnormal thyroid function
- Tingling, burning, numbness or weakness, possibly in arms, legs, hands and feet
- Vomiting

#### **UNCOMMON**: greater than or equal to 1 in 1,000 people to less than 1 in 100 people

- Abnormally excessive sweating involving the arms, legs, hands and feet, underarms, and face, usually unrelated to body temperature or exercise
- Bronchitis: inflammation of the lining of bronchial tubes, which carry air to and from the lungs
- Damage to the protective covering of the nerves in the brain and spinal cord
- Decreased secretion of hormones produced by adrenal glands
- Decreased thyroid stimulating hormone a lab test result associated with abnormal thyroid function
- Dehydration
- Diabetes: a disease that results in too much sugar in the blood
- Dry eye
- Erythema multiforme: a skin disorder that is considered to be an allergic reaction to medicine or an infection. Symptoms may include symmetrical, red, raised skin areas that can appear all over the body, more noticeable on the fingers and toes. These patches often look like "targets" (dark circles with purple-grey centers)
- Flu like symptoms (which may include fever, chills, cough, sore throat, runny or stuffy nose, muscle or body aches · headaches, feeling tired)
- Hair loss
- Heart rate increased

- Heart rhythm abnormal
- High blood pressure
- Hives
- Inflammation of the eye
- Inflammation of the kidney
- Inflammation of the liver
- Inflammation of the pancreas
- Inflammation of the pituitary gland
- Inflammation of the stomach
- Inflammation of the thyroid gland
- Kidney function failure, kidney disease
- Low blood pressure
- Low white blood cell counts (neutropenia): these put you at higher risk for infection
- Pemphigoid: blistering of the skin or mouth caused by the immune system attacking healthy tissue
- Psoriasis characterized by patches of abnormal, scaly skin
- Sarcoidosis a disease involving abnormal collections of inflammatory cells (granulomas) in organs such as lungs, skin, and lymph nodes
- Respiratory failure: a condition in which not enough oxygen passes from your lungs into your blood, or when your lungs cannot properly remove carbon dioxide
- Trouble falling and/or staying asleep (insomnia)
- Underactive function of the pituitary gland situated at the base of the brain
- Upper respiratory tract infection: a common viral / bacterial infection that affects the nose, throat, and airways
- Vision blurred

#### **RARE**: greater than or equal to 1 in 10,000 people to less than 1 in 1,000

- Autoimmune hemolytic anemia: a malfunction of the immune system that produces autoantibodies, which attack red blood cells as if they were foreign substances to the body
- Cranial nerve disorder can cause pain, tingling, numbness, weakness, or paralysis of the face including the eyes
- Diabetes complications resulting in excess blood acids
- Disease caused by the body's immune system attacking healthy organs
- Double vision
- Drug induced liver injury
- Guillain-Barre syndrome, an autoimmune disorder associated with progressive muscle weakness or paralysis
- Hemophagocytic lymphohistiocytosis (HLH) syndrome: a disease that may affect your body's defense system, called the immune system. Certain white blood cells may attack other blood cells. These abnormal blood cells collect in your spleen and liver, causing these organs to enlarge. The symptoms may include fever, rash, and low blood cell counts
- Histiocytic necrotizing lymphadenitis or Kikuchi lymphadenitis: disorder of the lymph nodes which causes the lymph nodes to become enlarged, inflamed and painful,

commonly affecting lymph nodes of the neck and possibly associated with fever or muscle and joint pains

- Inflammation of blood vessels (vasculitis)
- Inflammation of the brain, potentially life-threatening or fatal
- Inflammation of the heart
- Inflammation of the lining of the brain and spinal cord
- Lung infiltrates, associated with infection or inflammation
- Muscle inflammation
- Myasthenic syndrome neurologic syndrome characterized by muscle weakness including myasthenia gravis, a nerve disease that may cause weakness of eye, face, breathing, and swallowing muscles.
- Pericarditis: a swelling and irritation of the thin saclike membrane surrounding the heart (pericardium)
- Polymyalgia rheumatica a serious condition that causes inflammation of the lining of the arteries characterized by muscle pain and stiffness especially in the shoulders but can neck or hips.
- Rhabdomyolysis muscle fiber released into the blood stream which could damage your kidneys
- Rosacea acne-like skin condition resulting in redness of face
- Rupture of the intestine hole in the intestine
- Severe allergic reaction may include but not limited to high grade fever, rash, swelling and pain
- Stevens Johnson syndrome- a serious, potentially life threatening reaction of the skin and mucous membranes, resulting in blistering and shedding of skin
- Toxic epidermal necrolysis a potentially fatal disease characterized by blistering and peeling of the top layer of skin resembling a severe burn

The following events have been identified during post-approval use of nivolumab. Because reports are voluntary from a population of unknown size, an estimate of frequency cannot be made.

- Graft-versus-host-disease: a condition that occurs when donor bone marrow or stem cells attack the recipient
- Solid organ transplant rejection
- Vogt-Koyanagi-Harada (VKH) disease: a disease that may affect several parts of the body, including the eyes, ears, nervous system, and skin. The symptoms may include eye swelling, pain and/or blurred vision; hearing loss, ringing in the ears; and /or loss of skin color

<u>Immune System Disorders:</u> Nivolumab may cause your immune system to attack normal organs and cause side effects in many parts of the body. You should tell your study doctor or study nurse right away about any new symptoms you experience while receiving nivolumab.

Complications, including fatal events, have occurred in people who received allogeneic hematopoietic stem cell transplantation (HSCT) before or after nivolumab.

MCC #:20575

Complications, including rejection, have also been reported in people who have received an organ or tissue transplant. Study treatment with nivolumab may increase the risk of rejection of the organ or tissue transplant.

**Lung Inflammation (pneumonitis):** It is possible that nivolumab may cause inflammation of the tissues of the lung. This adverse effect has been reported infrequently in people receiving nivolumab. While many people with x-ray or CT abnormalities have not developed any symptoms, some people have developed mild to severe symptoms and in rare cases, death has occurred as a result of their lung inflammation. Signs and symptoms of lung inflammation may include:

- Difficulty breathing
- · Pain or discomfort while breathing
- Chest pain
- Cough
- Shortness of breath
- Increased rate of breathing
- Fever
- Low blood oxygen levels
- Fatigue

Your study doctor and study nurse will watch you closely for changes in your ability to breathe and for other signs or symptoms that might show you are developing this type of lung inflammation and will perform regular tests including physical exams, measurement of oxygen levels through non-invasive testing (for example, pulse oximeter), blood tests, chest x-rays and/or CT scans.

# Please inform your study doctor or study nurse <u>AT ONCE</u> if you experience any of the following:

- Any new or increased shortness of breath
- Any new or increased chest pain
- · Any new or increased pain/difficulty while breathing
- Any new or increased cough or any significant change in your type of cough; for example, any new or increased mucous or blood in your cough
- Any change in the amount of oxygen you require
- Any fever, fatigue, or other symptoms that occur at the same time as any changes to your breathing or other lung symptoms

If you start to develop symptoms, your study doctor will ask you to return to the clinic for additional tests, which could include a physical exam, measurement of oxygen levels, blood tests, chest x-rays, and/or CT scans. You will be monitored very closely for changes in your overall lung symptoms, monitoring may require hospitalization. You may require specific treatment in order to control pneumonitis. You may also be seen by a special doctor called a pulmonologist, who has special training to be an expert in how your lungs work.

MCC #:20575

Prolonged treatment with medicines that suppress inflammation, sometimes needed to manage the side effects of nivolumab study treatment, may lower your body's ability to fight off certain infections (for example, opportunistic infections). These infections may require treatment with antibiotic or antifungal medications and may be fatal.

#### Other Information and Possible Side Effects

Experience in people receiving GM-CSF protein (a protein that is produced by CG0070) suggests that people dosed with CG0070 could experience shortness of breath, dizziness, development of fluid leakage into the body cavities, and low blood pressure.

Treatment with high levels of GM-CSF may cause your immune system to react to GM-CSF and neutralize (reduce the effect) your body's natural GM-CSF proteins.

#### **ALLERGIC REACTION**

Occasionally, people have allergic reactions to drugs which may require medical treatment. A severe allergic reaction could be life-threatening. Examples of an allergic reaction include:

- Rash
- Shortness of breath
- Wheezing
- Difficulty breathing
- Sudden drop in blood pressure
- Swelling around the mouth, throat, or eye
- Fast pulse
- Sweating

You should get immediate medical help and contact the study doctor if you have any of these or any other side effects during the study.

## IS THERE ANY RISK TO YOUR UNBORN CHILDREN IF YOU TAKE PART IN THIS STUDY?

CG0070, DDM, and nivolumab may have adverse effects on a fetus in utero. Furthermore, it is not known if CG0070, DDM, or nivolumab have adverse effects on the composition of sperm. Taking these study medications may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study.

Nivolumab has been studied in laboratory and animal experiments to see if it causes problems with pregnancy or birth defects. In this case, we do not have enough information to determine if it could cause problems for a pregnancy or developing baby. However, even when the results are all normal it is still not possible to say that nothing bad will happen when a woman gets pregnant while she or her sexual partner is taking nivolumab.

MCC #:20575

#### FOR WOMEN:

If you are pregnant, you cannot participate in this study, because there may be risks to you and your unborn baby that are currently unforeseeable; risks that we do not know about yet. Breastfeeding (nursing) mothers will not be included in this study, since it is not known whether the study drugs in this study will be passed on to the baby in mother's milk. If you are currently breastfeeding and wish to continue breastfeeding, your study doctor may recommend another treatment.

If you are a female of childbearing potential, you will be given a pregnancy test before beginning any study drug. If you become pregnant while on this study, the study drug will be stopped immediately, and the pregnancy will be followed until conclusion.

Tell the study doctor right away if:

- You are pregnant
- You become pregnant
- You are planning to become pregnant
- You are breastfeeding

There may be risks to your unborn children that we don't know about ahead of time; they are unforeseeable.

If you take part in this study, you must use an effective birth control method as discussed with your study doctor. If you are a woman who can become pregnant you must use contraception during any sexual activity from the day of study drug initiation (or 14 days before the initiation of study medication for oral contraception) throughout the study period for up to 150 days after the last study treatment of CG0070, DDM, or nivolumab, whichever is later. No birth control requirements apply to postmenopausal women, those diagnosed with a congenital or acquired condition that prevents child-bearing, and those who had a hysterectomy and/or bilateral oophorectomy (removal of your womb and/or ovaries), bilateral salpingectomy (removal of your ovaries tubes) or bilateral tubal ligation/occlusion (also known as tubal sterilization or having your tubes tied or blocked), at least 6 weeks prior to Screening.

Examples of birth control methods include:

- Oral birth control pills
- Birth control patch
- Implanted (injectable contraceptive hormones or mechanical products such as intrauterine device)
- Barrier methods (such as: diaphragm, condoms, or spermicides)
- Tubal ligation or partner vasectomy
- Abstinence (no sexual intercourse)

You should discuss the method of birth control which is best for you to use both during study treatment and for a period of time after study treatment.

MCC #:20575

You should tell your study doctor immediately if you become pregnant or if your partner becomes pregnant. Women who become pregnant during the study will have to stop receiving the study drugs. The study doctor or study staff may ask for information about the pregnancy and the birth of the baby. If your partner becomes pregnant, she will be asked to sign and date a separate consent form to allow the study staff to collect information about the pregnancy, its outcome, and the health of the child after birth. The study doctor or study staff may share this information with the sponsor and Advarra IRB (a group of people who review research studies to protect the rights and welfare of research participants).

#### **Barrier Method**

It is not yet known of CG0070 can spread from person to person during sexual activity. Therefore, in addition to the contraception requirements above, a barrier method of contraception described above must be used from the start of CG0070 study treatment for up to 6 weeks after each CG0070 study treatment. This requirement applies to all participants regardless of age, gender, or ability to have a child.

# IF I AM TAKING MY REGULAR MEDICATION, WHAT ARE THE RISKS?

Taking other medications in combination with CG0070 and nivolumab may produce or worsen side effects of either study treatment when taken alone.

You will be asked at every visit to provide the names of any other medications you are taking or stopped during the study period. You should not take any other medications without first talking with your study doctor so that care can be taken to avoid combinations of medications that may be harmful to you. This includes prescription medications and over-the-counter medications, vitamins, herbal supplements, traditional medicines, and alcohol or recreational drugs

# COULD I HAVE ANY OTHER PROBLEMS WITH MY HEALTH IF I DO THIS RESEARCH STUDY?

It is possible that you could have problems and side effects of CG0070 and Nivolumab that nobody knows about yet, which include your condition getting worse or even death. If the study doctor learns any new information about study drugs that might change your mind about continuing in the study, the study doctor or study staff will tell you about it. The study doctor will also tell you if new treatments become available for your condition.

It is possible that taking, receiving, using CG0070 and Nivolumab with your regular medications or supplements may change how CG0070 and Nivolumab, your regular medications, or your regular supplements work. It is very important that you tell the study doctor about all medications or supplements you are taking during the study.

# WHAT ARE THE RISKS OF GIVING BLOOD FOR THIS STUDY?

Risks associated with drawing blood from your arm include momentary discomfort and/or bruising. Infection, excess bleeding, clotting, or fainting are also possible, although unlikely.

MCC #:20575

#### WHAT ARE THE RISKS OF HAVING A BIOPSY DONE FOR THIS STUDY?

## **Tumor Biopsy**

Risks of a tumor biopsy are localized bleeding at the needle injection site or from the surgical incision, pain, inflammation, swelling, and infection. The bleeding may cause discomfort and bruising. In rare circumstances (less than 1%), this bleeding may be severe enough to require further care. If you have a history of excessive bleeding, or if you are receiving medication that might increase your risk of bleeding (such as aspirin or blood thinners), you must notify the study doctor before the procedure. Infection of the surgical site may require treatment with antibiotics.

Any complications arising from the biopsy may be treated with observation, additional medications, or in some cases, additional surgery. The study doctor will discuss the specific risks of the biopsy with you at the time of the procedure.

#### WHAT ARE THE RISKS OF OTHER INVASIVE STUDY PROCEDURES?

#### **Urinary Catheterization**

Urinary Catheterization is a procedure where a flexible soft tube called a catheter is put into your bladder through your urethra, which allows urine to drain from the bladder. It is also used to inject liquids used for treatment and diagnosis of bladder conditions. You may feel pain and discomfort, bladder spasm which is quite common when the bladder tries to pass out the balloon section of the catheter. Rarely, bleeding can occur during the procedure due to trauma or injury. Urinary Tract Infection is the most common and can occur for some people.

#### **Intravesical Instillation (IVE Instillation)**

With intravesical therapy, the liquid drug is put right into your bladder. The study drug is given through a soft catheter that is put into your bladder through your urethra, which is the tube that leads from the bladder and transports and drains urine outside the body. The drug stays in your bladder for up to 1 hour. You may feel uncomfortable or pressure, irritation, a burning feeling in the bladder, and blood in the urine.

# Transurethral Resection of Bladder Tumor (TURBT)

It is a procedure in which the bladder tumor is removed from the bladder wall. It is performed completely with a scope that is inserted through the urethra into the bladder, you will be given an anesthesia medication before the procedure. During the procedure, the scope with a special cutting instrument is inserted through the natural channel into the bladder and then the tumor is removed.

You may feel burning sensation and some mild discomfort when urinating for several days. It is also common to have a change in the force of the urinary stream for several days and perhaps even 1–2 weeks.

Bleeding is also very common after this procedure. In the immediate hours after the procedure, there is often blood left over from the procedure that inevitably will color the urine bright red.

You may also be passing out some small clots during this time period. Usually, this bleeding will clear in 1–2 days. It is also very common for people to experience a small episode of repeat bleeding 1–2 weeks following his/her procedure. Typically, this is a small healing scab that is released from the urinary tract 1–2 weeks after the healing process has begun. This may be associated with a small amount of bleeding that should be self-limited.

If you start to have a temperature of 101 degrees or greater fever or if they begin passing clots that are larger than 1 inch in diameter, please contact your study doctor immediately.

As mentioned above, many people will have cherry colored urine, but may also experience darker burgundy-colored urine and at times brown-colored urine. The color of urine typically is determined by how long a time has passed since the bleeding began. If there is a significant amount of bleeding, you may require further examination or evaluation as it is usually associated with the passing of large clots as above.

#### Radical cystectomy, extended pelvic lymph node dissection

In this operation, the bladder, the prostate, the seminal vesicles (sperm sacs), and, if necessary, the urethra are removed. The ureters (which drain urine from the kidneys to the bladder) may be connected to a section of intestine that is connected to the surface of your abdomen at an opening called a urostomy or connected to a section of intestine formed into a "neobladder" which drains urine out of your urethra. Your surgeon will discuss the options with you. Risks include impotence for men and discomfort/difficulty with sexual intercourse for women, inability to father children for men, bleeding, infection, vitamin deficiency, diarrhea from a shorted intestine, bowel and/or urine leakage, and rectal injury. More specific risks to your specific procedure will be explained to you by your surgeon and you will be provided a separate surgical informed consent form for this procedure.

#### MRI

Magnetic resonance imaging (MRI) uses a magnet and radio waves to make diagnostic medical images of the body. There have been no ill effects reported from exposure to the magnetism or radio waves used in this test. However, it is possible that harmful effects could be recognized in the future. A known risk is that the magnet could attract certain kinds of metal. Therefore, we will carefully ask you about metal within your body, including medical implants, devices such as pacemakers and internal defibrillators, or certain dyes found in tattoos. We will also keep the examining room locked so that no one carrying metal objects can enter while you are in the scanner.

If there is any question about potentially hazardous metal within your body, you will not undergo the MRI. This may exclude you from participation in this research study. The MRI involves entering a large room in which a magnet is present. You will be placed on a narrow bed and then slid into a small tunnel approximately 6 feet in length and 25 inches in diameter. You will be asked to lie still for about one hour on this bed. You will hear a loud machine-like noise. You may be asked to have a harmless monitoring device applied during the MRI. During the MRI, you can have voice contact and physical contact with someone in attendance if you desire. Let the study doctor know if you have a fear of enclosed spaces.

MCC #:20575

#### CT Scan

Computed Tomography (CT) is a way to make x-ray images of the inside of the body. The CT scanner is a doughnut-shaped machine that uses x-rays to create computer pictures that show structures inside your body more clearly than regular x-ray pictures. During the procedure, a technologist will take you into the CT scan room where you will lie down on the table (usually on your back) inside of the CT machine. You should get comfortable because it is very important that you not move during certain parts of the test.

CT examinations differ depending on the part of your body being studied. For example, if your abdomen is being studied, a series of pictures will be taken from your lower chest to your lower pelvis. During the study, you will be asked to hold your breath so that the pictures will not be blurred. The machine will make some noise, and the table will move during the scan. Also, you may receive signals from the technologist or from the machine about your breathing. Before or during the study, you may be given an injection of a contrast liquid (dye) in your vein to allow the radiologist to obtain clearer images of your organs. This dye may cause you to get a metallic taste in your mouth and to feel warm. Rarely, it causes nausea and vomiting. The dye can also cause damage to kidneys, which may lead to kidney failure. This is a concern if you have poor kidney function. Rarely, the dye can cause a life threatening reaction. If you have any discomfort during the test or after the injection, be sure to tell the technologist.

#### **ALTERNATIVE TREATMENT:**

You do not have to be in this study to get help for the type of cancer you have. The study doctor will talk to you about other things you can do for this type of cancer, including the important risks and benefits.

Some other things you might do are:

- Use other approved chemotherapy regimens that do not include cisplatin
- Upfront radical cystectomy
- Use other investigational treatments
- Get supportive care or hospice care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Hospice care tries to keep you as active and comfortable as possible
- Choose to have no further treatment.

#### WHAT IF I GET HURT OR SICK WHILE I AM IN THIS STUDY?

# If you need emergency care:

 Call 911 or go to your nearest emergency room right away. Moffitt Cancer Center does not have an emergency room or the facilities to provide emergency care.

# If you do NOT need emergency care:

Call or go to your regular doctor. It is important that you tell your regular doctor that you
are participating in a research study. If possible, take a copy of this consent form with
you when you go.

MCC #:20575

If you experience a side effect or a change in the way that you feel, call the study doctor at the telephone number listed on the first page of this form.

By signing and dating this informed consent and research authorization form, you have not given up any legal rights to seek compensation for injuries from the sponsor.

#### MOFFITT CANCER CENTER INJURY STATEMENT

If you believe you have been injured as a result of your participation in this study or if you have questions about your rights as a person who is taking part in a research study, you may call the Moffitt Cancer Center Risk Manager at 813-745-7882. Moffitt Cancer Center and its investigators have made no provision for monetary compensation in the event of physical illness or injury resulting from this study. Likewise, Moffitt Cancer Center and its investigators have made no provision for payment of lost wages, disability, or discomfort in the event of physical illness or injury resulting from this study. Florida law (Statute 768.28) limits the liability of Moffitt Cancer Center. This statute provides that damages are available only to the extent that negligent conduct of a Moffitt Cancer Center employee caused your injuries, and are limited by law.

#### **WILL I GET PAID?**

You will not get paid for being in this study. You will not be reimbursed for expenses for travel and/or lodging while taking part in this study.

# INVESTIGATOR CONFLICT OF INTEREST STATEMENT

Roger Li, M.D., a person involved with this study, has received and may receive consultant and/or speaker fees from CG Oncology, Inc. fka Cold Genesys, a sponsor and/or supplier of drug for this study. This study has been carefully reviewed to help assure that the professional judgment of the Moffitt Cancer Center doctors and staff will not be compromised. The study will be monitored for your safety and for the proper analysis of data. Any questions you might have about this will be answered by the Moffitt Cancer Center Compliance Office at (813) 745-1869.

# WHILE YOU ARE IN THE STUDY, YOU MUST:

- Follow the instructions you are given.
- Come to the study center for all visits with the study doctor.
- Give correct and accurate information about your medical history and current medical condition.
- Tell the study doctor about any health problems you have during the study.
- Tell the study doctor about any new medicine or drug you take during the study.
- Not take any other drugs or remedies unless the study doctor has approved them beforehand. This includes prescription drugs and over the counter medicine (including vitamins and herbal remedies) that you buy without a prescription.

- Not participate in other medical research studies.
- Not get pregnant or cause your partner to become pregnant.
- Tell the study doctor or study staff if you want to stop being in the study at any time.

#### DO I HAVE TO REMAIN ON THIS STUDY ONCE I JOIN?

If you want to stop being in the study, tell the study doctor or study staff and return all unused study drug and study materials.

If you stop being in the study early, the study doctor or study staff may ask you some questions about being in the study. To help you leave the study safely, the study doctor may ask you to participate in more tests or return for a final study visit.

# ARE THERE REASONS THE STUDY DOCTOR OR SPONSOR MIGHT TAKE ME OUT OF THE STUDY LATER?

Even if you want to stay in the study, there may be reasons the study doctor or study staff will need to take you out of it. Your study doctor has the right to take you out of the study at any time with or without your agreement. Your participation may be ended without your consent for different reasons, including the following:

- If the study doctor believes, for any reason, that it is in your best interest.
- If at any time while you are taking the study drug the study doctor discovers that your disease has worsened.
- If you develop side effects that the study doctor considers unacceptable.
- If you refuse to take the study drug or return for follow-up as recommended by your study doctor, or do not follow the study doctor's instructions.
- If you refuse to have tests that are needed to determine whether the study drug is safe and effective.
- If you require treatment with drugs that are not allowed on this study.
- If other causes prevent you from continuing in this study.
- If the Sponsor decides to end the study.

#### **HOW WILL MY INFORMATION BE KEPT CONFIDENTIAL?**

We understand that information about you and your health is personal, and we are committed to protecting the privacy of that information. Because of this commitment and because of federal law, we must obtain your written authorization before we use or disclose your information for this study.

By signing and dating this form, you are permitting researchers at Moffitt Cancer Center to use personal health information for research purposes within its organized health care arrangements. You are also allowing the Moffitt Cancer Center to disclose your personal health information to outside organizations or individuals that participate in this study. We may publish what we find out from this study. If we do, we will not let anyone know your name. We will not publish anything that would directly let people know who you are.

Identifiers might be removed from your identifiable private information or identifiable biospecimens collected during this study and could then be used for future research studies or distributed to another investigator for future research studies without additional informed consent.

#### WHO WILL DISCLOSE, RECEIVE, AND/OR USE YOUR INFORMATION?

Your records are confidential and they will be kept in a secure environment and protected to the full extent of the law.

To do this research, the following people and/or organization(s) will be allowed to disclose, use, and receive your information, but they may only use and disclose the information to the other parties on this list, to you or your personal representative, or as permitted by law:

- Every research site for this study, including the Moffitt Cancer Center, and each site's study team, research staff and medical staff.
- Any person who provides services or oversight responsibilities in connection with this study.
- Every member of the Moffitt Cancer Center workforce who provides services in connection with this study.
- The person who is responsible for the study nationwide or worldwide (study chairperson).
- Any laboratories, individuals, and organizations that use your health information in connection with this study.
- Any sponsor of the study, including the following sponsors: Moffitt Cancer Center, CG Oncology
- Any federal, state, or local governmental agency that regulates the study (such as the U.S. Food and Drug Administration (FDA), Florida Department of Health (FDH) and Office for Human Research Protections (OHRP).
- Other government agencies in this or other countries.
- The designated Protocol Review and Monitoring Committees, Institutional Review Boards such as Advarra IRB, Privacy Boards, Data and Safety Monitoring Board and their related staff that have oversight responsibilities for this study.
- The National Cancer Institute in evaluating the ongoing research of the Moffitt Cancer Center as a Comprehensive Cancer Center.

The organizations and people listed above may employ or pay various consultants and companies to help them understand, analyze and conduct this study. All of these people may not be known now, but if you would like to have more specific information about this at any time during the study, you may ask the study doctor and your questions will be answered.

MCC #:20575

Moffitt Cancer Center cannot guarantee the privacy of your information, or block further use or distribution, after the information has left the Moffitt Cancer Center. Others listed above may further disclose your information, and it may no longer be covered by federal privacy regulations. If all information that does or can identify you is removed from your records, the remaining information will no longer be subject to this authorization and may be used or shared for other purposes. You might have the right to see and copy your health records related to this research. You might not be able to see or copy some of your records until after all participants finish the study. If it is necessary for your care, your records will be provided to you or your regular doctor.

#### WHAT INFORMATION WILL BE USED OR DISCLOSED?

By signing and dating below, you authorize the use and disclosure of your entire study record and any medical or other records held by Moffitt Cancer Center, including, but not limited to, HIV/AIDS, mental health, substance abuse or genetic information. The purpose for the uses and disclosures you are authorizing is to conduct the study explained to you during the informed consent and research authorization process and to ensure that the information relating to that study is available to all parties who may need it for research purposes.

Your authorization to use your health information will never expire unless and until you expressly revoke it in writing to the study doctor listed on the first page of this form.

Any data collected before your letter will continue to be used as necessary to preserve the integrity of the study, however no additional information will be collected after you withdraw your authorization.

You do not need to sign this form, but if you do not, you cannot participate in this study.

You will receive a signed and dated copy of this form.

#### WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study, please contact the Investigator at the telephone number listed on the first page of this consent document. If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, and/or concerns or complaints regarding this research study, contact:

Bv mail:

Study Participant Adviser Advarra IRB 6100 Merriweather Dr., Suite 600 Columbia, MD 21044

• or call **toll free**: 877-992-4724

• or by **email**: adviser@advarra.com

MCC #:20575

Please reference the following number when contacting the Study Participant Adviser: Pro00045614.

#### WHERE CAN I GET MORE INFORMATION?

You may call the National Cancer Institute's (NCI) Information Service at: 1-800-4-CANCER (1-800-422-6237).

Visit the NCI's Websites at:

- CancerTrials: comprehensive clinical trial information at: <a href="http://cancertrials.nci.nih.gov">http://cancertrials.nci.nih.gov</a>
- CancerNet: accurate cancer information including PDQ at: <a href="http://cancernet.nci.nih.gov">http://cancernet.nci.nih.gov</a>

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Information for Participants Receiving CG0070:

The study team will provide you with the instructions following after CG0070 and nivolumab study treatment. CG0070 is a weakened adenovirus that is capable of selective replicates in cancer cells. You should adhere to the following recommendation, as a precaution:

- Practice good hand hygiene with soap and warm water or with hand rubs containing at least 60% alcohol.
- Avoid direct physical contact with children less than 12 months of age and the individuals potentially at higher risk of exposure as defined above for at least 14 days after the last treatment.
- Do not share eating utensils or other objects that have come into contact with body fluids for at least 14 days after study treatment.
- After each CG0070 study treatment, participants are to abstain from intimate physical contact with others, including kissing and any sexual contact activity for at least 14 days after study treatment.
- A barrier method of contraception or other adequate means of contraception is to be used during study treatment and for 6 weeks after the last study treatment with CG0070; and used for 5 months (women or 7 months (men) after the last study treatment with nivolumab
- Dispose of contaminated materials such as urinary catheters, gloves, bandages, and dressing in a sealed container or sealed bag in the regular trash or return to the clinic for biohazard bag disposal.
- Clothing, bedding, and towels can be laundered in hot water with laundry detergent and approximately one cup of undiluted house bleach per wash load, for at least 14 days after study treatment
- For the first 14 days after receiving CG0070, you and your close contacts/family should avoid direct contact with your urine. Undiluted household bleach should be used to clean any urine spills and for routine disinfection of the toilet.

If you develop a *febrile respiratory illness, ocular (eye) disease,* or *diarrhea* potentially related to CG0070 study treatment, you should adhere to the following recommendation for at least 14 days after the study treatment:

- Avoid direct physical contact with any potentially contaminated material (for example, urine-soiled clothing or bedding). If patient care is necessary (for example, use of urinary catheters), gloves should be worn, and hands should be washed afterward with soap and warm water or hand rub containing at least 60% alcohol.
- Avoid touching other parts of your body (for example, eyes, nose, or other areas) after coughing, going to the bathroom or handling any other potentially contaminated material (for example, after changing a dressing or urinary catheter).
- If the symptoms of respiratory illness present:
  - Wear a mask when around other people
  - o Do not share items such as toothbrushes, eating utensils, etc.
- Dispose of contaminated materials (such as, urinary catheter, gloves, gauze, bandages) in a sealed container or sealed bag in regular trash or return to the clinic for biohazard bag disposal.
- Fabrics (such as, clothing, sheets, towels) can be laundered in hot water with detergent adding bleach to inactivate the virus (one cup per wash load).

I authorize Blood and Tissue for Future Research as described in section 'HOW WILL MY BLOOD/TISSUE SAMPLES BE USED?

| ☐ Yes | Participant Signature | | Date |
|---|---|---|---|
| □ No | Participant Signature | | Date |
| STATEM | ENT OF CONSENT AND AUTHOR | RIZATION | |
| for the pu | ad this form and its contents were e<br>urposes listed above. All of my que<br>signed and dated copy of this form | stions were answered to m | _ |
| Printed N | lame of Participant | | |
| Signature | e of Participant | <br>Date | |

STATEMENT OF PERSON OBTAINING INFORMED CONSENT / RESEARCH AUTHORIZATION

I attest that the participant named above had enough time to consider this information, had an opportunity to ask questions, and voluntarily agreed to be in this study.

| Printed Name of Person Explaining Consent | | |
|-------------------------------------------|----------|------|
| Signature of Person Explaining Consent | <br>Date | Time |

Sponsor Protocol Number: CORE-002